CLINICAL TRIAL: NCT02209311
Title: Effectiveness and Safety of Method of Maxilla Alveolar Process Reconstruction Using Tissue Engineered Construction Based on a Synthetic Tricalcium Phosphate and Autologous Multipotent Mesenchymal Stromal Cells Obtained From Oral Mucosa
Brief Title: Effectiveness and Safety of Method of Maxilla Alveolar Process Reconstruction Using Synthetic Tricalcium Phosphate and Autologous MMSCs
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Central Clinical Hospital w/Outpatient Health Center of Business Administration for the President of Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RU-CCH-06-01-14
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Partially Edentulous Maxilla; Alveolar Bone Atrophy; Alveolar Bone Loss
Keywords: Alveolar Bone Loss; Alveolar Bone Atrophy; Dental Implantation; Bone Tissue Reconstruction; Sinus Lift; Autologous Multipotent Mesenchymal Stem Cell; Autologous MMSCs; Synthetic Tricalcium Phosphate; Tissue Engineered Construction; Oral Mucosa
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tissue engineered construction implantation (Experimental)
  Interventions: Procedure: Oral mucosa biopsy; Procedure: Sinus lift with implantation of tissue engineered construction; Device: Dental implant

INTERVENTIONS:
Procedure: Oral mucosa biopsy
Procedure: Sinus lift with implantation of tissue engineered construction
Device: Dental implant

SUMMARY:
Autologous MMSCs will be isolated from oral mucosa biopsy sample and expanded in vitro.Tissue engineered construction will be created using synthetic tricalcium phosphate and autologous MMSCs. Patients will undergo sinus lift procedure with implantation of created tissue-engineered construction. This is a single arm study with no control. All patients receive cell therapy.

DETAILED DESCRIPTION:
Patients with verified diagnosis partially edentulous maxilla and alveolar bone atrophy will undergo oral mucosa biopsy and autologous MMSCs will be derived and expanded in vitro during 3-4 weeks. After that tissue engineered construction will be created using synthetic tricalcium phosphate and autologous MMSCs. Patients will undergo sinus lift procedure with implantation of created tissue-engineered construction. Six months later patients will undergo dental implant installation. Biopsy of bone tissue at the site of sinus lift will be performed as a part of dental implant installation with subsequent histological analysis of bone specimen.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous maxilla
* Height of the bone tissue in the area of reconstruction 1 - 5 mm according to results of cone-beam computed tomography
* Minimal height of the augmentation - 8 mm
* Volume of bone tissue deficiency of the alveolar process of the maxilla 3 - 5 cm3
* Implant installation scheduled to be at least 6 months after sinus-lift operation
* Patient is familiar with Participant information sheet
* Patient signed informed consent form

Non-inclusion Criteria:

* Chronic and acute ear, nose and throat diseases, including maxillary sinusitis, foreign bodies in the maxillary sinus, odontogenic and not odontogenic maxillary sinus cyst
* Medical history of surgery on maxillary sinuses during preceding 6 months prior to implantation of tissue engineered construction
* Progressive somatic disease (clinically significant diseases of the cardiovascular, hematopoietic or endocrine system, systemic diseases, immunopathological states)
* Patients with malignant tumors including postoperative period, patients receiving chemotherapy and/or radiotherapy
* Any conditions limiting compliance (dementia, neuropsychiatric disease, drug and alcohol abuse etc.)
* Significant weight loss (> 10% of body weight in the previous year) of unknown etiology
* Patient prescribed for any medications with proven effect on bone metabolism
* Diabetes mellitus, disorders of thyroid and parathyroid glands
* Clinically significant abnormalities in results of laboratory tests
* Participation in other clinical trials (or administration of investigational drugs) during 3 months prior inclusion

Exclusion Criteria:

* Patient's refusal from the further participation in trial
* Patient's refusal from compliance with the requirements of contraception during the participation in research
* Plaque index (PI)> 15%
* Sulcus bleeding index (SBI) > 10%
* Chronic kidney disease IV - V stages (creatinine clearance < 30 mL/min estimated by Cockroft-Gault formula)
* Confirmed syphilis, HIV, hepatitis B or C infections

Dropout Criteria:

* Perforation of the Schneider's membrane more than 5 mm on the stage of the sinus-lift operation
* Pregnancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-10 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Number of serious adverse events (SAEs) and serious adverse reactions (SARs) | 1 week after treatment

SECONDARY OUTCOMES:
Quality of life monitoring | up to 24 weeks after treatment
  Quality of life estimated by validated questionnaire: the Short Form (36) Health Survey (SF-36).
Changes in bone tissue volume | up to 24 weeks after treatment
  Changes in volume and density of bone tissue at the site of manipulation and newly formed bone micro-architecture assessed by cone beam CT (morphometrical analysis using Hounsfield unit measurements)
Correlation of morphometrical analysis using cone beam CT scan with absolute value of the newly formed bone | 24 weeks after treatment
  Biopsy of bone tissue at the site of sinus lift will be performed as a part of dental implant installation. Bone sample will be evaluated histologically: absolute value of the newly formed bone will be calculated using histomorphometrical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Grigory Volozhin A Volozhin, MD, PhD, Principal Investigator — A.I. Evdokimov Moscow State Medical Stomatological University; Ilya I Eremin, MD, PhD, Principal Investigator — Federal State Budgetary Institution "Central Clinical Hospital with Outpatient Health Center" of the Business Administration for the President of the Russian Federation; Center for Biomedical Technologies
Locations (2):
- Russia (2):
  - Federal State Budgetary Institution "Central Clinical Hospital with Outpatient Health Center" of the Business Administration for the President of the Russian Federation; Center for Biomedical Technologies, Moscow
  - A.I. Evdokimov Moscow State Medical Stomatological University, Moscow